CLINICAL TRIAL: NCT04254692
Title: Randomized Controlled Trial Evaluating Liposomal Bupivacaine Following Abdominoplasty
Brief Title: Optimizing Recovery in Abdominoplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: division wide research suspension
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-1570; A539730 (Other: UW Madison); SMPH/SURGERY/DENTL-PLASTC SRGY (Other: UW Madison); Protocol Ver 2, 04/09/2021 (Other: UW Madison)
Record Dates: First submitted 2019-12-23; First posted 2020-02-05 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
Keywords: abdominoplasty; enhanced recovery after surgery; Liposomal bupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine (Active Comparator): Participants in this study arm will receive intraoperative injection of Liposomal Bupivacaine mixed with Bupivacaine to the abdominal wall.
  Interventions: Drug: Liposomal bupivacaine
- Bupivacaine (Other): Participants in this study arm will receive intraoperative injection of bupivacaine without Liposomal bupivacaine to the abdominal wall.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Liposomal bupivacaine — Participants in the intervention group will receive intraoperative injection of Liposomal bupivacaine mixed with Bupivacaine to the abdominal wall.
  Arms: Liposomal Bupivacaine
Other: Standard of care — Participants in the standard of care group will receive intraoperative injection of bupivacaine only to the abdominal wall
  Arms: Bupivacaine

SUMMARY:
The overall purpose of this study is to evaluate the analgesic efficacy of liposomal bupivacaine in optimizing pain control, minimizing the risk of postoperative nausea and vomiting (PONV), and improving recovery after abdominoplasty. This will be done by comparing intraoperative abdominal wall and incisional injection of bupivacaine to bupivacaine plus liposomal bupivacaine in 46 participants 18 years and older undergoing elective abdominoplasty. This will be studied using pain assessments, validated surveys, medication logs and review of medical records.

DETAILED DESCRIPTION:
Postoperative pain, nausea, and vomiting can be frustrating sequelae of elective surgery. Poorly managed postoperative pain can lead to increased opioid use, increased postoperative nausea and vomiting (PONV), delayed return to work and usual activities, unplanned hospital admissions, surgical complications, and patient dissatisfaction. In light of the growing opioid epidemic in the United States, any intervention that potentially minimizes opioid use may have meaningful individual and societal impact. Despite the use of multiple techniques for managing postoperative pain in abdominoplasty patients, pain control continues to be a challenge for this patient population.

One technique commonly employed to improve pain control is the use of abdominal wall and incisional injection of local anesthetic agents to block the sensory nerves supplying the anterior abdominal wall and abdominal incisions in order to decrease sensation and pain in the abdomen in the setting of abdominoplasty surgery. Local anesthetic often used in this procedure is bupivacaine (Marcaine) ± epinephrine. However, in 2012, a liposomal bupivacaine suspension (Exparel; Pacira BioSciences, Inc, San Diego, California) was introduced as a longer-acting local anesthetic used for management of postoperative pain. At the University of Wisconsin, patients undergoing abdominoplasty routinely receive intraoperative injection of local anesthetic to the abdominal wall and abdominal incisions, using bupivacaine as the local anesthetic, along with standard multimodal perioperative pain management including cool compresses, non-steroidal anti-inflammatories (NSAIDs), acetaminophen, and opioids.

The overall purpose of this study is to evaluate the analgesic efficacy of liposomal bupivacaine in optimizing pain control, minimizing the risk of PONV, and improving recovery after abdominoplasty. This will be done by comparing intraoperative abdominal wall and incisional injection of bupivacaine to bupivacaine plus liposomal bupivacaine in patients undergoing abdominoplasty. This will be studied using pain assessments, validated surveys, medication logs and review of medical records.

ELIGIBILITY:
Inclusion Criteria:

* Medically cleared to undergo elective surgery (including associated anesthesia) at UW Madison Surgery Center (MSC).

Exclusion Criteria:

* Pregnant or breast-feeding women
* Incarcerated women or men
* Individuals unable to give consent due to another condition such as impaired decision-making capacity.
* Men or women who take opioid pain medications on a regular basis prior to surgery
* Men or women with a history of opioid abuse and/or dependence
* Participants with a history of bleeding disorders precluding safe abdominoplasty
* Participants on anticoagulation therapy who have not held their anticoagulation as recommended by their surgeon or anesthesiologist
* Participants not medically cleared for surgery at Madison Surgery Center. This would include participants with sepsis/bacteremia, significant valvular disorders or heart conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venkat Rao, MD, MBA, Principal Investigator — University of Wisconsin Hospitals and Clinics
Locations (2):
- United States (2):
  - University of Wisconsin Madison Surgery Center, Madison, Wisconsin
  - University of Wisconsin Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data collection occurred from 1/5/2021 to 1/21/2021
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Bupivacaine | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 54 [54 to 54] | 35 [35 to 35] | 45.1 [35 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
Body Mass Index (BMI) [Number; unit: kilograms per meter squared] | 25.8 | 19.1 | 22.5

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use at 24 Hours
Description: Amount of opioids used postoperatively, measured in morphine equivalents
Time Frame: 24 hours postoperatively
Measure: Number; unit: morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 1 | 1
morphine milligram equivalents | 0 | 15

2. Secondary Outcome: Quality of Recovery-40 (QOR-40) Score
Description: The QOR-40 is a 40 item survey about the quality of recovery with a total possible range of scores from 40 to 200 where the higher the score the higher quality the recovery.
Time Frame: 24 hours postoperatively
Measure: Number; unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 1 | 1
score on a scale | 161 | 168

3. Secondary Outcome: Pain Score Postoperative Day 1 (POD 1)
Description: The pain survey is scored on a 0-10 scale where 0 is no pain and 10 is the worst possible pain.
Time Frame: 24 hours postoperatively
Measure: Number; unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 1 | 1
score on a scale | 6.5 | 8

4. Secondary Outcome: Pain Score 1 Week Postop
Description: The pain survey is scored on a 0-10 scale where 0 is no pain and 10 is the worst possible pain.
Time Frame: 1 week postoperatively
Measure: Number; unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 1 | 1
score on a scale | 2 | 1

5. Secondary Outcome: Opioid Use at 1 Week
Description: total opioid used, measure in morphine equivalents
Time Frame: 1 week postoperatively
Measure: Number; unit: morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 1 | 1
morphine milligram equivalents | 0 | 0

6. Secondary Outcome: Antiemetic Use POD 1
Description: total antiemetic used
Time Frame: 24 hours postoperatively
Measure: Number; unit: antiemetic doses
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 1 | 1
antiemetic doses | 0 | 0

7. Secondary Outcome: Antiemetic Use 1 Week
Description: total antiemetic used
Time Frame: 1 week postoperatively
Measure: Number; unit: antiemetic doses
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 1 | 1
antiemetic doses | 0 | 0

8. Secondary Outcome: Number of Participants With Postoperative Nausea and Vomiting
Time Frame: 24 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Postoperative Complications
Time Frame: 1 week postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 1 week post op
Arm/Group | Liposomal Bupivacaine | Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
study terminated early, not powered for meaningful results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT04254692/Prot_SAP_000.pdf